CLINICAL TRIAL: NCT02362165
Title: A Phase 3 Trial Comparing Cyclophosphamide,Bortezomib,and Dexamethasone (CyBorD) and Bortezomib,Doxorubicin,and Dexamethasone (PAD) in the Treatment of Newly Diagnosed Multiple Myeloma
Brief Title: CyBorD vs. PAD in the Treatment of Newly Diagnosed Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xia Zhongjun, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-MM-308
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; cyclophosphamide; bortezomib; doxorubicin; peripheral neuropathy
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases | interventions — Cyclophosphamide; Bortezomib; Dexamethasone; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CyBorD regimen (Experimental): this arm will receive cyclophosphamide (500mg/d,once-weekly),bortezomib(1.3mg/㎡，once-weekly,subcutaneous injection), and dexamethasone (40mg/d,once-weekly)(CyBorD) as induction therapy.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone
- PAD regimen (Active Comparator): this arm will receive bortezomib(1.3mg/㎡，once-weekly,subcutaneous injection), dexamethasone (40mg/d,once-weekly), and doxorubicin (9mg/㎡，d1-4)(PAD) as induction therapy.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — 500mg/d,once-weekly,per oral.
  Other Names: endoxan
  Arms: CyBorD regimen
Drug: Bortezomib — 1.3mg/㎡,once-weekly,subcutaneous injection
  Other Names: velcade
Drug: Dexamethasone — 40mg/d,once-weekly,per oral
Drug: Doxorubicin — 9mg/㎡,d1-4
  Other Names: adriamycin
  Arms: PAD regimen

SUMMARY:
Bortezomib-based triple-drug combination has greatly improved the response rate of multiple myeloma patients. Bortezomib,doxorubicin,and dexamethasone (PAD) is commonly used in clinical practice.Recent studies have found that cyclophosphamide, bortezomib,and dexamethasone (CyBorD)seems better than PAD in efficacy. However, there is no randomized phase 3 trial comparing these two regimens in the treatment of newly diagnosed multiple myeloma patients.In this study, the investigators will compare the efficacy and safety of these two regimens using once-weekly subcutaneous injection of bortezomib.

DETAILED DESCRIPTION:
Bortezomib-based triple-drug combination has greatly improved the response rate of multiple myeloma patients. Bortezomib,doxorubicin,and dexamethasone (PAD) is commonly used in clinical practice. Recent studies have found that cyclophosphamide, bortezomib,and dexamethasone (CyBorD)seems better than PAD in efficacy. However, there is no randomized phase 3 trial comparing these two regimens in the treatment of newly diagnosed multiple myeloma patients. Moreover, studies have found that subcutaneous injection of bortezomib can decrease the incidence rate of peripheral neuropathy induced by bortezomib, however, most center use twice-weekly administration of bortezomib. According to our experience, once-weekly subcutaneous injection of bortezomib can further decrease the incidence rate of peripheral neuropathy without compromising the efficacy. Thus, in this phase 3 trial, the investigators will compare the efficacy and safety of these two regimens using once-weekly subcutaneous injection of bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of multiple myeloma
* Eastern Cooperative Oncology Group (ECOG) status 0-3,
* Estimated survival time > 3 months
* Acceptable liver function (bilirubin<2.5×ULN, Alanine transaminase (ALT) or Aspartate Aminotransferase (AST)<2.5×ULN)
* No history of other malignancies
* No previous treatments including chemotherapy, radiotherapy, targeted therapy or stem cell transplantation
* No other serious diseases which conflict with the treatment in the present trial
* No concurrent treatments that conflict with the treatments in the present trial
* Voluntary participation and signed the informed consent.

Exclusion Criteria:

* The patients had the conditions below: clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), symptomatic coronary artery heart disease requiring medication;
* The patients participated in other clinical trials within the 30 days before enrollment or who are participating in other clinical studies
* The patients with neuropathy
* The patients with mentally ill / unable to obtain informed consent
* The patients with drug addiction, alcohol abuse which affects the long-term evaluation of test results
* The patients in pregnancy, lactation and women of childbearing age who do not want to take contraceptive measures subjects
* The patients with a history of allergy to test drug
* The patients not suitable to participate in the investigator judged by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
At least very good partial response rate (according to the criteria IMWG) after four cycles of induction therapy | date from randomization to 1 month after completion of 4 cycles of induction therapy (up to 6 months)
  compare the Response assessment in both arms: the Very good partial response rate (according to the criteria IMWG) achieved with four courses of CyBorD with with that achieved with four courses of PAD

SECONDARY OUTCOMES:
complete response rate(according to the criteria IMWG) after four cycles of induction therapy | date from randomization to 1 month after completion of 4 cycles of induction therapy (up to 6 months)
  compare the Response assessment in both arms: the complete response rate (according to the criteria IMWG) achieved with four courses of CyBorD with with that achieved with four courses of PAD
At least partial response rate (according to the criteria IMWG) after four cycles of induction therapy | date from randomization to 1 month after completion of 4 cycles of induction therapy (up to 6 months)
  compare the Response assessment in both arms: the at least partial response rate (CR+VGPR+PR) (according to the criteria IMWG) achieved with four courses of CyBorD with with that achieved with four courses of PAD

CONTACTS AND LOCATIONS:
Overall Officials: Zhongjun Xia, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen university cancer center, Guangzhou, Guangdong, China